CLINICAL TRIAL: NCT02935725
Title: A Phase 1, Single-centre, Double-blind, Placebocontrolled Crossover Study to Assess the pharmacoMRI Effects of AUT00206 in Healthy Male Participants
Brief Title: A Study to Assess the pharmacoMRI Effects of AUT00206 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autifony Therapeutics Limited (Industry)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AUT021206; 2016-000216-14 (EudraCT Number)
Record Dates: First submitted 2016-08-15; First posted 2016-10-17 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose AUT00206 800 mg + Ketamine (Experimental): Low dose AUT00206 (800 mg) + ketamine
  Interventions: Drug: Low dose AUT00206 800mg; Drug: Ketamine
- High dose AUT00206 2000 mg + Ketamine (Experimental): High dose AUT00206 (2000 mg) + ketamine
  Interventions: Drug: High dose AUT00206 2000 mg; Drug: Ketamine
- Placebo + Ketamine (Placebo Comparator): Placebo + ketamine
  Interventions: Drug: Placebo; Drug: Ketamine
- Placebo + Saline (Placebo Comparator): Placebo + saline
  Interventions: Drug: Placebo; Other: Saline

INTERVENTIONS:
Drug: Low dose AUT00206 800mg
  Arms: Low dose AUT00206 800 mg + Ketamine
Drug: High dose AUT00206 2000 mg
  Arms: High dose AUT00206 2000 mg + Ketamine
Drug: Placebo
  Arms: Placebo + Ketamine; Placebo + Saline
Drug: Ketamine
  Arms: High dose AUT00206 2000 mg + Ketamine; Low dose AUT00206 800 mg + Ketamine; Placebo + Ketamine
Other: Saline
  Arms: Placebo + Saline

SUMMARY:
A Phase 1, Single-centre, Double-blind, Placebo controlled Crossover Study to Assess the pharmacoMRI Effects of AUT00206 in Healthy Male Participants

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 to 45 years, inclusive at Visit 1.
* Healthy on the basis of medical history, psychiatric history, physical examination, vital signs, 12-lead electrocardiogram (ECG), haematology, blood chemistry and urinalysis within 6 weeks of Visit 2.
* Right-handed.
* Not a regular smoker (maximum 5 cigarettes per week or equivalent).

Exclusion Criteria:

* History of, or current condition of, migraine headaches or has undergone operations to the head.
* History of significant claustrophobia.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Significant difference in BOLD phMRI signals after dosing with AUT00206 vs placebo | 15 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bill Deakin, Prof, Principal Investigator — University of Manchester
Locations (1):
- University Of Manchester, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be made publicly available on completion of the trial.